CLINICAL TRIAL: NCT03793621
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BI 730357 in Japanese Healthy Male Subjects (Double-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: This Study is Done in Healthy Japanese Volunteers. It Looks at How Different Doses of BI 730357 Are Taken up in the Body and How Well They Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1407-0015
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 730357 (Experimental)
  Interventions: Drug: BI 730357
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 730357 — single rising oral dose
  Arms: BI 730357
Drug: Placebo — single rising oral dose
  Arms: Placebo

SUMMARY:
The main objective of this trial is to investigate the safety and tolerability of BI 730357 in Japanese healthy male subjects following oral administration of single rising doses.

Secondary objectives are the explorations of the pharmacokinetic(s) (PK), including dose proportionality as well as investigation of linearity of BI 730357 after single dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR), Respiratory Rate (RR), body temperature), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Japanese ethnicity, according to the following criteria:

  -- born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
* Age of 20 to 45 years (inclusive) at screening
* Body Mass Index (BMI) of 18.5 to 25.0 kg/m2 (inclusive) at screening
* Signed and dated written informed consent in accordance with International Council for Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male subject who agree to minimize the risk of female partners becoming pregnant by fulfilling any of the following criteria starting from participation to this trial and until 90 days after the trial completion:

  * Use of adequate contraception, e.g., any of the following methods plus condom:

    --- combined oral contraceptives, intrauterine device.
  * Vasectomised (vasectomy at least 1 year prior to enrolment)
  * Surgical sterilised (including hysterectomy) of the subject's female partner

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic BP outside the range of 90 to 140 mmHg, diastolic BP outside the range of 50 to 90 mmHg, or PR outside the range of 45 to 90 beats per minute (bpm) at screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance at screening
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the Central Nervous System (CNS) (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders, including but not limited to mood disorders and any history of suicidality
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including human immunodeficiency virus (HIV), viral hepatitis, syphilis and/or tuberculosis
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days or 5 half-lives, whichever is longer, prior to administration of trial medication, if that might reasonably influence the results of the trial (including potential for QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Previous exposure to BI 730357
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day for males)
* Drug abuse or positive drug screening
* Whole blood donation of more than 200 mL within 30 days or 400 mL within 12 weeks, or plasmapheresis and platelet apheresis within 2 weeks prior to administration of trial medication, or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 mseconds) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigation of safety and tolerability of BI730357 in healthy subjects following oral administration of single rising doses of 50, 100, and 200mg. The trial was designed as double-blind, randomised within dose group, and placebo-controlled within parallel dose group.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be entered to trial treatment if any of the specific entry criteria were not met.
Groups:
- Placebo: Placebo film-coated tablet (1 for 50 milligram (mg) group, 1 for 100 mg group, 2 for 200 mg group), administered as single oral dose with ~240 milliliter of water after an overnight fast of at least 10 hours. Subjects receiving placebo were equally distributed across dose groups.
- 50 mg BI 730357 Single Dose: 1 film-coated tablet (50 milligram) of BI 730357, administered as single oral dose with ~240 milliliter of water after an overnight fast of at least 10 hours.
- 100 mg BI 730357 Single Dose: 1 film-coated tablet (100 milligram) of BI 730357, administered as single oral dose with ~240 milliliter of water after an overnight fast of at least 10 hours.
- 200 mg BI 730357 Single Dose: 2 film-coated tablets (100 milligram each) of BI 730357, administered as single oral dose with ~240 milliliter of water after an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | Placebo | 50 mg BI 730357 Single Dose | 100 mg BI 730357 Single Dose | 200 mg BI 730357 Single Dose
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS), which included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg BI 730357 Single Dose | 100 mg BI 730357 Single Dose | 200 mg BI 730357 Single Dose | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.7 (7.6) | 22.2 (1.8) | 26.8 (7.3) | 32.8 (7.3) | 27.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 6 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-related Adverse Events
Description: Number of participants with trial drug-related adverse events.
Time Frame: Up to 7 days after drug administration.
Population: Treated Set (TS):
  All subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subject received.
Measure: Number; unit: Participants
Arm/Group | Placebo | 50 mg BI 730357 Single Dose | 100 mg BI 730357 Single Dose | 200 mg BI 730357 Single Dose
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 730357 in Plasma Over the Time Interval From 0 Extrapolated to Infinity
Description: Area under the concentration-time curve of BI 730357 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Within 3 hours before drug administration and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 34, 48, 72, 96 and 168 hours after drug administration.
Population: Pharmacokinetics analysis set (PKS): All subjects in the treated set (TS) who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Only participants with non-missing results are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*Nanomoles per Litre (h*nmol/L)
Arm/Group | 50 mg BI 730357 Single Dose | 100 mg BI 730357 Single Dose | 200 mg BI 730357 Single Dose
Number analyzed (Participants) | 5 | 6 | 4
Hours*Nanomoles per Litre (h*nmol/L) | 7160 (14.3) | 13000 (48.6) | 13200 (53.1)

3. Secondary Outcome: Maximum Measured Concentration of BI 730357 in Plasma
Description: Maximum measured concentration of BI 730357 in plasma (Cmax).
Time Frame: as for outcome 2
Population: Pharmacokinetics analysis set (PKS): All subjects in the treated set (TS) who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per Litre (nmol/L)
Arm/Group | 50 mg BI 730357 Single Dose | 100 mg BI 730357 Single Dose | 200 mg BI 730357 Single Dose
Number analyzed (Participants) | 6 | 6 | 6
Nanomoles per Litre (nmol/L) | 346 (23.0) | 451 (34.8) | 515 (48.2)

ADVERSE EVENTS:
Time Frame: [Serious and Other Adverse Events]: Up to 7 days after drug administration. [All-cause mortality]: From drug administration until end of trial, up to 13 days.
Description: Adverse events are reported based on treated set (TS). This set included all subjects who were randomized and treated with at least 1 dose of trial drug. The TS was used for safety analyses.
Arm/Group | Placebo | 50 mg BI 730357 Single Dose | 100 mg BI 730357 Single Dose | 200 mg BI 730357 Single Dose | Total
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 1/6 | 1/24
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | 50 mg BI 730357 Single Dose (N=6) | 100 mg BI 730357 Single Dose (N=6) | 200 mg BI 730357 Single Dose (N=6) | Total (N=24)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT03793621/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT03793621/SAP_001.pdf